CLINICAL TRIAL: NCT06224140
Title: Heparin-Free Chronic HemoDialysis Assessment
Acronym: HepFreeHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCAPHM21_0424_HEPFREEHD
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heparin Anticoagulation (Active Comparator)
  Interventions: Procedure: Heparin Anticoagulation
- Regional Anticoagulation Procedure (RAP) (Experimental)
  Interventions: Procedure: Regional Anticoagulation Procedure (RAP)

INTERVENTIONS:
Procedure: Heparin Anticoagulation — Conventional dialysis with heparin as anticoagulant treatment
  Arms: Heparin Anticoagulation
Procedure: Regional Anticoagulation Procedure (RAP) — Dialysis without heparin as anticoagulant but based on the use of a calcium-free dialysis bath. Calcium is then restored by reinjection of a 10% calcium chloride solution.
  Arms: Regional Anticoagulation Procedure (RAP)

SUMMARY:
Intermittent hemodialysis is a complex technique which requires careful monitoring of anticoagulation levels to prevent clotting and reduce the risk of bleeding complications. Dialysis patients often exhibit hypercoagulable tendencies due to uremic state, turbulent blood flows in dialysis procedures, and thrombogenic exposure to artificial surfaces of dialysis tubing. Patients with ESRD may experience both dialyzer clotting and excessive bleeding, so individualized heparin dosing and periodic adjustments are necessary to ensure adequate anticoagulation during hemodialysis. The ideal anticoagulant should prevent thrombosis while minimizing the risk of intra- and interdialytic bleeding. The use of heparin carries risks such as worsening of osteoporosis and dyslipidemia, allergic reactions like pruritus, and the potential for life-threatening heparin-induced thrombocytopenia (HIT) for which avoidance of heparin is necessary during dialysis.Heparin, in both its unfractionated heparin (UFH) and low molecular weight heparin (LMWH) forms, is the most commonly used anticoagulant, though evidence comparing their efficacy and risk of bleeding remains inconclusive. End-stage renal disease (ESRD) patients, who are already at higher risk of serious bleeding, may benefit from regional anticoagulation (RA) techniques, as they typically receive around 600,000 IU of heparin per year. The investigators performed routinely a simplified regional anticoagulation procedure (RAP) using a constant calcium re-injection rate over the time to avoid hypocalcemia. This procedure eliminates the need for citrate infusion and calcium monitoring, and reduces nurse workload in a chronic dialysis unit. The investigators compared 21 chronic dialysis patients with 198 RA and 195 heparin sessions, where each patient acted as their own control. None of them were on VKA during the RA sessions, 62% were on single anti-platelet therapy and 14% were on dual anti-platelet therapy. The dialysis session success rate was 94% in the RA group and 97% in the heparin group, with no significant differences (p=0.22). The circuit loss rate was 1.5% per RA session and 0.5% per heparin session (p=0.23), and the early blood restitution rate was 3% and 1.5% (p=0.50) in the RA and heparin groups, respectively

Hypothesis: RAP can be as effective as systemic anticoagulation with heparin for intermittent dialysis in chronic hemodialysis patients, with the potential to reduce the rate of hemorrhagic events

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or more
* Patients with end-stage renal disease (ESRD) under intermittent hemodialysis, for more than 3 months prior to screening and with a dialysis duration prescription of at least 4 hours
* Effective anticoagulation either by UFH or by LMWH of the dialysis session defined by the absence of circuit loss in the last 3 months.
* Dialysis adequacy defined by a mean Kt/V ≥1.2.
* Calcemia within the normal range at inclusion (2.2 to 2.6 mmol/L) (based on the results of the last monthly blood test)
* Subject affiliated to or beneficiary of a social security system.
* Subject having signed written informed consent.

Exclusion Criteria:

* Dysfunctional vascular access at the screening
* Unipunction of the AVF
* Patient treated by hemofiltration or hemodiafiltration procedure
* Current anticoagulation treatment
* Patient treated by digitalizing drugs
* Patient treated by thiazide diuretics
* Patient with hypercalcemia and/or hypercalciuria
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Active hemorrhage
* High bleeding risk defined by the following situations: recent bleeding of less than 7 days, recent post-operative period of less than 7 days, recent head trauma of less than 7 days, recent ischemic stroke of less than 7 days, uremic pericarditis.
* Body weight < 45 kg and > 140 kg at screening.
* Known allergy to citrate
* Hospitalization at the screening for all other causes apart from dialysis
* Moribund status (defined by the expectation of death in less than three months).
* Liver failure (to prevent citrate liver toxicity) based on the results of the last monthly or quarterly blood test
* Ongoing participation in a concurrent interventional study in dialysis or with anti-coagulation therapy
* Pregnancy (declarative) or breastfeeding and all the other categories of people with special protection according to the French Code de la Santé Publique (CSP): patients under legal supervision, patients hospitalized without consent, patients admitted in social or sanitary structures for care and not research, and patients in emergency situations
* Patients unable to give an informed consent or unwilling to participate in the study.
* Heparin-coated membrane in current dialysis prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the non-inferiority of the regional anticoagulation procedure compared to heparin anticoagulation on the dialysis sessions success three times per week | 6 months
  The primary endpoint will be the rate of dialysis sessions success over 6 months between two therapeutic strategies:
  * Regional anticoagulation procedure (RAP)
  * Heparin anticoagulation

SECONDARY OUTCOMES:
Compare between the groups clinical Impact at each dialyses session on bypass loss | 6 months
  Rate of bypass loss
Compare between the groups clinical Impact at each dialyses session on early bypass restitution | 6 months
  Rate of early bypass restitution (defined as a restitution 30 minutes or more before the end of the prescribed time)
Compare between the groups clinical Impact at each dialyses session on dialysis duration | 6 months
  Mean difference of dialysis duration over 6 month between the groups
Compare between the groups clinical Impact at each dialyses session on fistula compression time extended more than 10 minutes | 6 months
  Rate of fistula compression time extended more than 10 minutes after a dialysis session
Compare between the groups clinical Impact during the total duration of the study on incidence of hemorrhagic events | 6 months
  Incidence rate of hemorrhagic events
Compare between the groups clinical Impact during the total duration of the study on dialysis adequacy | 6 months
  Time average-dialysis adequacy difference defined by the average kt/v over 6 months
Compare between the groups clinical Impact during the total duration of the study on relative effects on phosphocalcic balance | 6 months
  Mean difference at months +6 and time-average evolution over 6 month for calcium, phosphor, bone-specific alkaline phosphatase and parathyroid hormone concentration between the groups
Compare between the groups clinical Impact during the total duration of the study on incidence of Hyperparthyroidism | 6 months
  Rate of hyperparathyroidism defined par PTH > 9N at month +6
Compare between the groups clinical Impact during the total duration of the study on incidence of non-hemorrhagic heparin-related complications | 6 months
  Rate of non-hemorrhagic heparin-related complications:
  1. In the heparin group: heparin-induced thrombocytopenia,
  2. Between the groups: hyperkalemia, hypertriglyceridemia, hypersensitivity reactions, pruritus at months +6
Compare between the groups clinical Impact during the total duration of the study on incidence of cardiovascular-related mortality and major cardiovascular events (MACE) | 6 months
  Incidence rate of MACE at months +6
Compare between the groups clinical Impact during the total duration of the study on global mortality | 6 months
  All-cause mortality rate at month +6
Compare between the groups the tolerance of per-dialytic hypotension | 6 months
  Rate of per-dialytic hypotension over 6 months
Compare between the groups the tolerance of adverse events | 6 months
  Rate of adverse events over 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Conception, Marseille, Bouches du Rhône, France

IPD SHARING:
Plan to Share IPD: No